CLINICAL TRIAL: NCT05918835
Title: Deciphering the Neural Mechanisms of Restrictive Eating in Anorexia Nervosa Using Repetitive Transcranial Magnetic Stimulation
Brief Title: Effects of rTMS on Food Choice in Anorexia Nervosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Eating Disorders Association (Other); Global Foundation for Eating Disorders (Unknown)
Responsible Party: Principal Investigator, Alexandra F Muratore, PhD, Assistant Professor of Clinical Medical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: #8338; 1K23MH128530 (NIH)
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: Repetitive Transcranial Magnetic Stimulation; Anorexia Nervosa; Restrictive Eating; Feeding and Eating Disorders
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High-frequency repetitive transcranial magnetic stimulation (HF-rTMS) (Experimental): Target: Region of right DLPFC with greatest resting-state functional connectivity to dorsal striatum (individualized functional target) Protocol: 10 pulses/sec, 4s trains, 120% MT, 3000 pulses/session
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation (active rTMS)
- Sham repetitive transcranial magnetic stimulation (sham rTMS) (Sham Comparator): Target: Region of right DLPFC with greatest resting-state functional connectivity to dorsal striatum (individualized functional target) Protocol: same as HF-rTMS, with sham coil
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (sham rTMS)

INTERVENTIONS:
Device: High-frequency repetitive transcranial magnetic stimulation (active rTMS) — HF-rTMS is applied with a figure-of-8 coil using the Magstim TMS System. Participants receive one administration of HF-rTMS, delivered to the region of the right dorsolateral prefrontal cortex (DLPFC) with greatest resting-state functional connectivity to the dorsal striatum (individualized per participant). HF-rTMS is delivered at a frequency of 10 Hz for approximately 37 minutes (3000 total pulses).
  Other Names: Magstim TMS System active coil; High-frequency rTMS; Repetitive Transcranial Magnetic Stimulation
  Arms: High-frequency repetitive transcranial magnetic stimulation (HF-rTMS)
Device: Sham repetitive transcranial magnetic stimulation (sham rTMS) — Sham rTMS is applied with a figure-of-8 sham coil using the Magstim TMS System, which is identical to the active coil, replicates the sounds of HF-rTMS, and is designed to mimic sensations of HF-rTMS. Participants receive one administration of sham rTMS, delivered to the region of the right dorsolateral prefrontal cortex (DLPFC) with greatest resting-state functional connectivity to the dorsal striatum (individualized per participant). Sham rTMS is delivered for approximately 37 minutes (3000 total pulses).
  Other Names: Magstim TMS System sham coil; Sham rTMS
  Arms: Sham repetitive transcranial magnetic stimulation (sham rTMS)

SUMMARY:
This study will examine the impact of high-frequency repetitive transcranial magnetic stimulation on food choice behavior and related neural activity.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a devastating illness with morbidity and mortality rates among the highest associated with any psychiatric disorder. Treatments for adults with AN have limited efficacy due to an inadequate understanding of the mechanisms underlying AN's core symptoms. The salient feature of AN is extreme restriction of food, particularly dietary fat intake, a behavior both highly resistant to change and central to relapse. Neuroimaging research of food restriction in AN has found that compared to healthy controls, patients with AN exhibit greater choice-related dorsal striatum activation and different connection strength within dorsal fronto-striatal circuits, suggesting that activity in this region and associated circuits may underlie maladaptive eating behavior. To confirm the significance of these brain regions in restrictive eating, this study will combine neuronavigation-guided high-frequency rTMS (HF-rTMS), individualized functional TMS targets, fMRI and a computerized food-choice task to test the effects of HF-rTMS on restrictive food choice and associated neural activity.

The study will utilize a double-blinded randomized parallel design: adult inpatients with AN will receive either HF-rTMS or sham to the DLPFC. We will compare group changes in brain and behavior to test whether activity in the dorsal striatum underlies restrictive eating behavior in AN and quantify the effects of HF-rTMS to the DLPFC on restrictive eating behavior. Our use of individualized TMS targets will enable us to identify whether resting-state functional connectivity predicts neural or behavioral response to HF-rTMS.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Diagnosis of Anorexia Nervosa
* Age 18-30 years
* Female
* Right-handed
* Body Mass Index (BMI) ≥ 16.0
* Voluntarily admitted to inpatient eating disorders unit at NYSPI
* Competent to provide informed consent
* English-speaking
* Medically stable

Exclusion Criteria:

* High risk of suicide
* Current substance use disorder or other co- morbid psychiatric condition requiring specialized treatment (e.g., psychosis)
* Diagnosis of major medical or neurological problem or taking medication that significantly increases risk for seizure or affects interpretation of findings (e.g., unstable hypertension, seizure disorder)
* Food restrictions (e.g., allergies) which impact greater than 30% of food choice task's choice options
* Indwelling ferromagnetic metallic object (e.g., pacemaker, pump), non- removable metal jewelry, medicinal patch or recent metallic ink tattoo
* History of seizure
* Diagnosis of epilepsy, stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, or parenchymal or leptomeningeal cancers
* Prior exposure to TMS
* Pregnancy
* Currently breast-feeding
* Significant claustrophobia
* Implanted devices or stimulators
* Hearing loss (e.g., currently undergoing treatment with ototoxic medications or those with cochlear implants)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Neural activity and functional connectivity during the food choice task | Baseline to post-treatment (approx. 1 week apart)
  Change in: food choice-related BOLD activity within the dorsal striatum, food choice-related functional Change in: connectivity between the dorsal striatum and dorsolateral prefrontal cortex
Restrictive eating behavior during the food choice task | Baseline to post-treatment (approx. 1 week apart)
  Change in: proportion of high-fat foods selected; proportion of trials in which participants had an opportunity to implement self-control; proportion of trials in which participants implemented self-control

SECONDARY OUTCOMES:
Predictors of HF-rTMS response | Baseline to post-treatment (approx. 1 week apart)
  Association between resting-state functional connectivity and: neural activity and functional connectivity during the food choice task (primary outcome #1); restrictive eating behavior during the food choice task (primary outcome #2)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra F Muratore, PhD, Principal Investigator — New York Sate Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No